CLINICAL TRIAL: NCT01519388
Title: Evaluation of Nasal Ventilation on Optimizing Swallowing in Ventilated Neuromuscular Patients
Brief Title: Evaluation of the Impact on Swallowing of Non Invasive Ventilation
Acronym: OPTIDEG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre d'Investigation Clinique et Technologique 805 (Other)
Collaborators: Adep Assistance (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2011-A00771-40
Record Dates: First submitted 2012-01-23; First posted 2012-01-26 (Estimated); Last update posted 2013-07-10 (Estimated); Status verified 2013-07

CONDITIONS: Neuromuscular Disorder; Respiratory Failure; Swallowing; Mechanical Ventilation
Keywords: Neuromuscular disorder; Respiratory failure; Swallowing; Mechanical ventilation
MeSH Terms: conditions — Neuromuscular Diseases; Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- neuromuscular patients (Experimental): Neuromuscular non invasively ventilated patients in stable at the time of the study
  Interventions: Other: Spontaneous breathing; Device: Elysée 150®

INTERVENTIONS:
Other: Spontaneous breathing — study of the swallowing of boluses of water and yogurt under spontaneous breathing
Device: Elysée 150® — Study of the swallowing of boluses of water and yogurt while under mechanical ventilation

SUMMARY:
Neuromuscular disorders can be associated with swallowing dysfunction secondary to a dysfunction of the airway muscles involved in swallowing. The investigators have shown that respiratory failure may contribute to swallowing dysfunction in patients with neuromuscular respiratory failure. Furthermore, although tracheostomy has been reported as impairing swallowing, the investigators have shown that when a tracheostomy is performed in neuromuscular patients, swallowing improves because it allows the patient to feed while ventilated.

The investigators now want to evaluate whether non invasive ventilation may have a beneficial impact on swallowing by making some adjustments to ensure a good synchronisation between ventilation and swallowing. This could allow avoiding the necessity of a tracheostomy or a gastrostomy due to swallowing dysfunction and/or malnutrition in neuromuscular patients.

Swallowing improvement under mechanical ventilation depends on improving the synchronisation between the patient and the ventilator during swallowing. For that purpose, the investigators developed a prototype ventilator able to temporarily suspend pressurisation under the patient's control so that when the patient needs to swallow under mechanical ventilation he may do so with an inadequate insufflation of the ventilator.

Our objective is to to demonstrate that swallowing is more adapted and easier under nasal noninvasive ventilation than during spontaneous breathing in neuromuscular patients requiring prolonged noninvasive ventilation.

In an open monocentric pilot study, the investigators will study 10 neuromuscular patients usually noninvasively ventilated. The patients will be their own control and their swallow will be studied during spontaneous breathing and under ventilation with the adapted ventilator while swallowing boluses of different volumes.

DETAILED DESCRIPTION:
Neuromuscular disorders can be associated with swallowing dysfunction secondary to a dysfunction of airway muscles involved in swallowing. We have shown that respiratory failure may also contribute to swallowing dysfunction and that, although tracheostomy has been reported as impairing swallowing, when a tracheostomy was performed in neuromuscular patients, swallowing was improved because it allowed the patient to feed while ventilated.

We now want to evaluate whether non invasive ventilation may have a beneficial impact on swallowing considering some adjustments to ensure a good synchronisation between ventilation and swallowing. This could allow avoiding the necessity of a tracheostomy or a gastrostomy due to swallowing dysfunction and/or malnutrition. Improving swallowing under mechanical ventilation depends on improving the synchronisation between the patient and the ventilator during swallowing. For that purpose, we developed a prototype ventilator able to temporarily suspend pressurisation under the patient's control so that when the patient needs to swallow under mechanical ventilation he may do so with an inadequate insufflation of the ventilator.

Our objective is to to demonstrate that swallowing is more adapted and easier under nasal noninvasive ventilation than during spontaneous breathing in neuromuscular patients requiring prolonged noninvasive ventilation.

In an open monocentric pilot study, we will study 10 neuromuscular patients usually noninvasively ventilated. The patients will be their own control and their swallow will be studied during spontaneous breathing and under ventilation with the adapted ventilator while swallowing boluses of different volumes. Swallowing will be evaluated by measuring swallowing duration, numbers of swallows required for a bolus, number of respiratory cycles required for the swallow of a bolus. Order ventilation mode and bolus volume will be randomized

ELIGIBILITY:
Inclusion criteria:

* Neurologic or Neuromuscular restrictive respiratory failure, excluding bulbar involvement
* Hospitalization in the home ventilation unit of the Raymond Poincaré Hospital
* day and night non invasive ventilation during >14hours/day
* respiratory autonomy of at least one hour of during the day
* Ventilation with an assisted and controled mode
* Adults ≥18 years
* Stable patient upon inclusion
* prior Medical examination
* Signed consent form

Exclusion Criteria:

* Unstable hemodynamics
* Respiratory decompensation
* Unable to cooperate
* Person under guardianship or trusteeship
* Pregnant women
* Refusal of study participation
* Non covered by the social security system

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-02; Primary Completion 2012-02 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
impact of non invasive ventilation on swallowing efficiency | 2 Hours
  Swallowing efficiency under non invasive ventilation will be evaluated by the duration of swallowing of bolus, number of swallow per bolus, number of respiratory cycles per swallowed bolus

SECONDARY OUTCOMES:
Swallow and respiration synchronisation | 2 Hours
  Number of swallows followed by expiration
Respiratory comfort | 2 Hours
  Evaluation of the respiratory comfort by the Borg dypnea scale

CONTACTS AND LOCATIONS:
Overall Officials: Helene PRIGENT, Md-PhD, Principal Investigator — Raymond Poincare Hospital - Garches - France; Frederic LOFASO, MD-PhD, Study Director — Raymond Poincare Hospital - Garches - France
Locations (1):
- Raymond Poincare Hospital, Garches, Garches, France

REFERENCES:
- [Background] Prigent H, Lejaille M, Terzi N, Annane D, Figere M, Orlikowski D, Lofaso F. Effect of a tracheostomy speaking valve on breathing-swallowing interaction. Intensive Care Med. 2012 Jan;38(1):85-90. doi: 10.1007/s00134-011-2417-8. Epub 2011 Nov 24. PMID 22113817
- [Background] Terzi N, Prigent H, Lejaille M, Falaize L, Annane D, Orlikowski D, Lofaso F. Impact of tracheostomy on swallowing performance in Duchenne muscular dystrophy. Neuromuscul Disord. 2010 Aug;20(8):493-8. doi: 10.1016/j.nmd.2010.05.009. Epub 2010 Jun 16. PMID 20558065
- [Background] Terzi N, Orlikowski D, Aegerter P, Lejaille M, Ruquet M, Zalcman G, Fermanian C, Raphael JC, Lofaso F. Breathing-swallowing interaction in neuromuscular patients: a physiological evaluation. Am J Respir Crit Care Med. 2007 Feb 1;175(3):269-76. doi: 10.1164/rccm.200608-1067OC. Epub 2006 Nov 16. PMID 17110642
- [Derived] Garguilo M, Lejaille M, Vaugier I, Orlikowski D, Terzi N, Lofaso F, Prigent H. Noninvasive Mechanical Ventilation Improves Breathing-Swallowing Interaction of Ventilator Dependent Neuromuscular Patients: A Prospective Crossover Study. PLoS One. 2016 Mar 3;11(3):e0148673. doi: 10.1371/journal.pone.0148673. eCollection 2016. PMID 26938617